CLINICAL TRIAL: NCT06900127
Title: The Effects Of Safe Swadding On Newborns' Oxygen Saturation And Comfort Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayse Sonay Turkmen, Prof.Dr (Other)
Responsible Party: Sponsor-Investigator, Ayse Sonay Turkmen, Prof.Dr, Prof. Dr., Karamanoğlu Mehmetbey University
Organization: Karamanoğlu Mehmetbey University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Safe Swaddling
Record Dates: First submitted 2025-03-14; First posted 2025-03-28 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Newborn; Fit; Safety Issues
Keywords: Safe Swaddling; Comfort; Saturation; Newborn

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe Swaddling (Experimental)
  Interventions: Behavioral: Safe Swaddling
- control group (No Intervention)

INTERVENTIONS:
Behavioral: Safe Swaddling — newborns will be wrapped with the safe wrapping method.
  Arms: Safe Swaddling

SUMMARY:
Objective: This study was conducted as a randomized controlled experimental study to determine the effects of safe swaddling on oxygen saturation and comfort in preterm newborns born between 30-36 weeks of gestation.

Methods: The sample of the study consisted of 70 newborns (Safe swaddling group =35, control group=35) hospitalized in the neonatal intensive care unit of a university hospital in Türkiye. The preterm newborns in the safe swaddling group were monitored by applying the safe swaddling method outside of care hours (12:00, 18:00, 24:00, 06:00), while those in the control group were followed in accordance with the hospital routines. An information form and a newborn comfort behavior scale were used as data collection tools. Descriptive statistics, chi-square, t test, Anova, analysis of variance in repeated measures, and Tukey forward analysis were used to evaluate the data.

DETAILED DESCRIPTION:
The population of the study consisted of preterm newborns receiving treatment in the Tertiary Neonatal Intensive Care Unit of X University Medical Faculty Hospital. Preterm babies between 30-36 weeks of gestation were included in the sample. The sample size of the study was accepted as type 1 error probability (α) 0.05 (95% confidence level) and type 2 error probability (β) 0.10 (80% power level), taking into account the known score in the G*Power 3.1.5 program. The sample size was determined as 32 for each group. However, since it was thought that there might be loss during the analysis, it was planned to reach 35 newborns for each group. As a result of the study, a total of 70 preterm newborns who met the inclusion criteria were reached.

Randomization The distribution of the newborns included in the study into groups was created by a statistician using codes obtained from a permutation-based computer program and stratified according to gestational age. The groups represented by the letters were determined at the beginning of the study using the closed opaque envelope method. As a result of the draw, it was decided that the letter A would represent the control group, and the letter B would represent the safe swaddling group. A single-participant blinding was applied in the study. A separate informed consent form was created and approved for each group. Thus, each newborn parent received information only about the intervention that would be applied to him/her. Randomization was followed according to the CONSORT 2010 diagram.

Hypotheses H1: Safe swaddling applied to preterm newborns has an effect on mean comfort scores.

H2: Safe swaddling applied to preterm newborns has an effect on oxygen saturation.

Data Collection Tools The study data were collected using the Information Form, Neonatal Comfort Behavior Scale (COMFORTneo), Neonatal Bedside Monitor, and Histogram Tracking Form.

Information form 10 questions containing introductory information in the information form (age, gender, delivery method, birth order, height and weight, etc.) consist of a question determining the status of special care and a newborn follow-up chart (daily oxygen saturation, comfort score, behavioral response status, and pain).

Newborn Comfort Behavior Scale (COMFORTneo) The scale is a Likert-type scale developed to assess the need for sedation and comfort, pain, and distress of newborns monitored in intensive care.

Neonatal bedside monitor The SpO2 data of the newborn taken with the bedside monitor were obtained from Philips IntelliVue MP40 model monitors in 24-hour periods. This monitor was preferred because it has a histogram feature. Data is stored in the monitor as 24-hour oxygen saturation trends.

Histogram tracking form In the Neonatal Intensive Care Unit, SpO2 monitoring is recorded via monitors and expressed as a percentage. The percentages of histogram data obtained through monitors are recorded. According to the histogram saturation evaluation results, preterm newborns received oxygen support as per clinical practice. The method of oxygen support given varies depending on the needs of the preterm newborn. Therefore, newborns whose 24-hour saturation trend is below 20% in the undesirable range (1-90%) in the histogram evaluation are considered hypoxia and therefore immediate intervention is required. Oxygen support is applied as NIMV (NCPAP, AIRVO, HF, LF, respectively) and free flow.

Data collection For the control group, safe swaddling was not applied, and routine hospital care and treatments were continued. The newborn's comfort assessment was made by two observers using the Neonatal Comfort Behavior Scale (COMFORTneo) every day at 10:00 during the data collection period. Histogram measurements were also taken by the researcher at 10:00 as a 24-hour oxygen saturation record. The newborn's height, weight, feeding frequency and amount were taken by the researcher every day at 10:00 during the data collection period and recorded on the data collection form. As for the safe swaddling group: safe swaddling was applied to the newborn by the researcher at the beginning of the study. Safe swaddling was applied after the newborn completed the 72nd hour after birth. The swaddle was removed only during care hours, for an average of 20 minutes. The newborn was then swaddled again by the same researcher. Since there are four care hours per day in the hospital routine, this total duration was accepted as 80 minutes. The newborn's comfort assessment was made by two observers using the Newborn Comfort Behavior Scale (COMFORTneo) every day at 10:00 during the data collection period. Histogram measurements were also taken by the researcher at 10:00 as a 24-hour oxygen saturation record. The newborn's height, weight, feeding frequency and amount were taken by the researcher every day at 10:00 during the data collection period and recorded on the data collection form.

Evaluation of Data The data obtained were evaluated in the computer environment using descriptive statistics (number, percentage, mean, standard deviation, min-max values), chi-square, t-test, Anova, analysis of variance in repeated measures, and Tukey advanced analysis in the SPSS 21 package program.

Ethical Aspects of the Study The study was carried out in accordance with the ethical principles at every stage. Before implementing the study, ethical permission was obtained from the Non-Interventional Research Ethics Committee of X University Faculty of Health Sciences (dated 31.03.2021, numbered 01-2021/05) and institutional permission was obtained from X University Medical Faculty Hospital (dated 25.06.2021 and numbered E-30292447-045.99-91265). Written consent was obtained from parents who met the criteria to be included in the study on a voluntary basis.

ELIGIBILITY:
Inclusion Criteria:

* The baby's gestational age to be between 30 weeks and 36 weeks,

  * The baby's birth weight to be 1250 grams or more,
  * The baby's oxygen requirement to be 40% or less,
  * The baby's to be between 4-28 days old,
  * The swaddling to be done by the same nurse,
  * Parents must agree to participate in the study.

Exclusion Criteria:

* • In our study, the babies were not followed up during the first 72 hours because of possible interventions such as giving them surfactant, exposing them to more invasive procedures, and taking heel blood resulting fluctuations in their vital signs.

  * The baby's having any kind of congenital anomalies.
  * There being a situation that prevents swaddling.

Criteria for dropping from the study while the study is ongoing

* When the baby loses his/her life,
* When the family gives up participating in the study,
* When the baby is intubated.

Ages: 1 Day to 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
comfort | once a day until discharged (up to 60 days) Min.=6 points, Max.=30 points
  comfort score averages
oxygen saturation | every day until discharge (up to 60 days)
  daily oxygen saturation averages

SECONDARY OUTCOMES:
NCPAP | every day until discharge (up to 60 days)
  Number of days receiving NCPAP
hospitalization | every day until discharge (up to 60 days)
  days of hospitalization

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ayşe Sonay Türkmen, Karaman
  - Karamanoglu Mehmetbey University, Karaman